CLINICAL TRIAL: NCT01828411
Title: Monitoring the Brain in On-pump Cardiovascular Surgery: The Role of Transpharyngeal Ultrasonography as a Non-invasive Adjunct to Assess Cerebral Perfusion
Brief Title: Cerebral Perfusion Monitoring With Transpharyngeal Ultrasonography
Acronym: TP-Echo
Status: Terminated | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 056/10
Record Dates: First submitted 2013-03-27; First posted 2013-04-10 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Cardiopulmonary Bypass
Keywords: Cardiac surgery; Echocardiography; Cerebral perfusion; Intraoperative period

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cardiopulmonary bypass group: Patients requiring normothermic (or mild hypothermic) cardiopulmonary bypass.
  Interventions: Device: Transpharyngeal ultrasonography; Device: Duplex sonography
- Hypothermic Cardiopulmonary Bypass Group: Patients requiring (deep) hypothermic cardiopulmonary bypass.
  Interventions: Device: Transpharyngeal ultrasonography; Device: Duplex sonography

INTERVENTIONS:
Device: Transpharyngeal ultrasonography — Transpharyngeal Dopplerultrasonography (Device: iE33 xMatrix Philips). Assessment of cerebral blood flow by detection of blood flow velocities in the extracranial carotid arteries.
Device: Duplex sonography — Assessment of cerebral blood flow by detection of blood flow velocities in the extracranial carotid and middle cerebral arteries during coronary artery bypass grafting.

SUMMARY:
This prospective observational pilot study investigates transpharyngeal ultrasonography (TPU) as an additional neuromonitoring strategy to assess cerebral perfusion during on-pump cardiovascular surgery.

In the first part of the study the investigators will investigate the feasibility of TPU for visualization of aortic arch branches including the innominate and the carotid arteries in twenty patients undergoing coronary artery bypass grafting with extracorporeal circulation (cohort 1.). In the second part the investigators plan to adopt the investigators previous experiences on TPU to a selected population of twelve patients undergoing ascending aortic and/or arch repair in deep hypothermic circulatory arrest (DHCA, cohort 2.). In contrast to cohort 1., patients in cohort 2. are exposed intraoperatively to intermittent cerebral perfusion stops or reductions due to surgical procedure, perfusion technique and their underlying disease (aortic dissection or aortic aneurysm).

The investigators hypothesize that cerebral perfusion monitoring using TPU as a non-invasive technique provides a simple and real-time adjunct to assess blood flow velocity in the extracranial cephalic vessels with Doppler ultrasound. Especially in aortic arch surgery with its inherent risk of cerebral hypoperfusion TPU might be a valuable adjunct to routine.

DETAILED DESCRIPTION:
Background

Cerebral hypo- or malperfusion during cardiovascular surgery can lead to grave consequences including transient cerebral ischemia or stroke impairing patient's daily life and affect surgical outcome. For this reason a multimodal neuromonitoring strategy using a variety of devices (evoked potentials, near-infrared spectroscopy, transcranial Doppler ultrasonography) with different technologies has been recommended by medical societies. These techniques have various limitations and cannot be used in all clinical situations. In contrast, transpharyngeal ultrasonography (TPU) represents a simple and readily available technique: the transesophageal echocardiography probe, routinely placed in most cardiac surgical patients for monitoring and assessment of surgical results, will be withdrawn into the upper esophagus making the visualization of supraaortic branches possible.

To date, there are several reports about imaging of aortic arch branches using TPU. The utility of this technique, however, for systematic cerebrovascular monitoring has not have been investigated so far.

Objective

The aim of this study is to investigate TPU as a cerebrovascular monitoring adjunct in two cohorts of on-pump cardiac surgery procedures. Clinical feasibility and diagnostic accuracy of antegrade carotid flow detection are compared to the established reference methods of Duplex sonography and transcranial Doppler ultrasound.

Methods

All patients receive anesthetic and surgical management according to institutional standards. Patient enrollment in the study occurs consecutively and unblinded for surgical procedure.

All patients receive TPU, Duplex sonography and transcranial Doppler examination after anesthesia induction preoperatively, during extracorporeal circulation and after weaning from cardiopulmonary bypass. In addition, the patients in cohort 2.(ascending aortic repair with DHCA) receive above mentioned noninvasive ultrasound / Doppler measurements also during the period of DHCA with and without antegrade cerebral perfusion.

Image acquisition and data extraction are conducted by different persons to avoid investigator-related bias.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Cardiopulmonary bypass procedure (normo-(group 1) or hypothermic (group 2))

Exclusion Criteria

* Contraindication for transesophageal echocardiography
* Carotid artery stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery at the University Hospital Bern.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-04; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
accuracy of cerebral flow velocity measurement | intraoperative phase, expected to be ca. 4 hours
  Cerebral blood flow velocity measurements will be performed using the pulsed wave Doppler technique. Doppler peak flow velocities (obtained at the same intraoperative phase and at the same time) will be compared between the different Doppler techniques.

SECONDARY OUTCOMES:
clinical feasibility | intraoperative phase, expected to be ca. 4 hours
  Clinical feasibility will be assessed by analyzing the accuracy of data concordance, i.e. location of cerebral blood vessel, blood flow velocity and cerebral vessel area between the different Doppler techniques. Data will be plotted using Bland-Altman analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Balthasar Eberle, Prof., MD., Study Chair — University Hospital Bern, Dep. of Anesthesiology and Pain therapy
Locations (1):
- Dep. of Anesthesiology and Pain therapy, Bern, Switzerland

REFERENCES:
- [Background] Bevilacqua S, Romagnoli S, Ciappi F, Ridolfi N, Codecasa R, Rostagno C, Sorbara C. Transpharyngeal ultrasonography for cannulation of the internal jugular vein. Anesthesiology. 2005 Apr;102(4):873-4. doi: 10.1097/00000542-200504000-00038. No abstract available. PMID 15791132
- [Background] Shimizu H, Matayoshi T, Morita M, Ueda T, Yozu R. Total arch replacement under flow monitoring during selective cerebral perfusion using a single pump. Ann Thorac Surg. 2013 Jan;95(1):29-34. doi: 10.1016/j.athoracsur.2012.08.007. Epub 2012 Oct 4. PMID 23040825
- [Background] Orihashi K, Matsuura Y, Sueda T, Watari M, Okada K, Sugawara Y, Ishii O. Aortic arch branches are no longer a blind zone for transesophageal echocardiography: a new eye for aortic surgeons. J Thorac Cardiovasc Surg. 2000 Sep;120(3):466-72. doi: 10.1067/mtc.2000.108289. PMID 10962406
- [Background] Nanda NC, Miller AP, Nekkanti R, Aaluri S. Transpharyngeal echocardiographic imaging of the right and left carotid arteries. Echocardiography. 2001 Nov;18(8):711-6. doi: 10.1046/j.1540-8175.2001.00711.x. PMID 11801216
- [Background] Immer FF, Moser B, Krahenbuhl ES, Englberger L, Stalder M, Eckstein FS, Carrel T. Arterial access through the right subclavian artery in surgery of the aortic arch improves neurologic outcome and mid-term quality of life. Ann Thorac Surg. 2008 May;85(5):1614-8; discussion 1618. doi: 10.1016/j.athoracsur.2007.11.027. PMID 18442549